CLINICAL TRIAL: NCT04639635
Title: Study of CNGB1 Retinitis Pigmentosa and Allied Hereditary Disorders
Brief Title: CNGB1 and Allied Disorders
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Michigan State University (Other); Moorfields Eye Hospital NHS Foundation Trust (Other); Universität Tübingen (Other); Wills Eye (Other); La Fondation Voir et Entendre (Unknown); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: AAAS1160
Record Dates: First submitted 2020-08-07; First posted 2020-11-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Retinitis Pigmentosa Associated With CNGB1 Mutations
Keywords: Retinitis Pigmentosa; CNGB1; Natural Progression
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, this is a natural history progression study — The objective is to better understand the disease process of CNGB1-RP so that we can develop clinical tests to measure the outcomes of treatment.

SUMMARY:
Mutations in the rod-expressed gene, cyclic nucleotide-gated channel beta subunit (CNGB1) and associated inborn errors in metabolism are causes of retinal disease that causes progressive loss of vision. Retinitis pigmentosa (RP) is a major cause of untreatable blindness associated with CNGB1 (CNGB1-RP). RP involves the death of photoreceptor cells that can be caused by mutations in a number of different genes. Treatment by gene therapy could prevent blindness in cases of inherited retinal dystrophies including RP. In the future RP due to mutations in CNGB1 may be treatable by gene therapy since this form of photoreceptor degeneration involves a slow loss of rod photoreceptor cells. This provides a wide window of opportunity for the identification of patients and initiation of treatment. Our efforts are directed toward developing gene therapy as a treatment. To this end, our objective is to better understand the disease process of CNGB1-RP and other allied inherited disorders so that we can develop clinical tests to measure the outcomes of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CNGB1-associated RP by study physician, who are trained retinal specialists in the university clinic
* Must be able to commit to 4 follow-up study visits (3 years)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are expected to present to the clinic at all age groups; enrollment of subjects <18 years of age will be obtained by informed consent in the company of a parent or legal guardian. There will also be no gender-or ethnic/racial specific inclusion criteria. The enrollment of non-English speaking subjects is not expected.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
We will be looking to identify what the best outcome measurements will be for CNGB1-RP in order to use these measurements in a future clinical trial. | 2 days, 1 time per year, for 3 years
  Both structural imaging and functional tests will be used to characterize the natural history progression of CNGB1-RP.
Medmont Dark Adapted Chromatic (DAC) Automated Perimeter | 1 time per year, for 3 years
Full-field ERG (ISCEV Protocol) | 1 time per year, for 3 years
Optical Coherence Tomography (OCT) | 1 time per year, for 3 years
Fundus Autofluorescence (FAF) | 1 time per year, for 3 years
Near-infrared fundus autofluorescence (NIR-AF) | 1 time per year, for 3 years
Quantitative Fundus Autofluorescence (qAF) | 1 time per year, for 3 years

SECONDARY OUTCOMES:
Best-corrected Visual Acuity (BCVA) | 1 time per year, for 3 years
Complete Ophthalmic Exam | 2 time per year, for 3 years
Color Fundus Photos | 1 time per year, for 3 years
MAIA Microperimetry | 1 time per year, for 3 years
  if available
NIDEK Microperimetry | 1 time per year, for 3 years
  if available
Goldman Kinetic Visual Field | 1 time per year, for 3 years
Light-adapted Static Perimetry | 1 time per year, for 3 years
Panel D-15 Colour Vision (desat.) | 1 time per year, for 3 years
Dark-adapted Chromatic Perimetry | 1 time per year, for 3 years
Full-field Stimulus Testing (FST) | 1 time per year, for 3 years
  Optional

OTHER OUTCOMES:
Demographics/medical history | 1 time only at baseline
Concomitant medications/adverse events | 1 time only at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Tsang, MD, PhD, Principal Investigator — Columbia University
Locations (6):
- United States (2):
  - Dr. Stephen H. Tsang, New York, New York
  - Wills Eye Hospital, Philadelphia, Pennsylvania
- Institut de la Vision/Centre de maladies rares du Centre Hospitalier National Ophtalmologique des Quinze-Vingts, Paris, France
- Germany (2):
  - Klinikum der Universität München University Eye Hospital, Ludwig-Maximilians-University (LMU) Munich, München, Bavaria
  - Eberhard Karls University Tubingen, Tübingen
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom